CLINICAL TRIAL: NCT05277727
Title: Impact of a Novel Marine Algae Supplement on the Inflammatory and Immune Response After High Intensity Exercise
Brief Title: Inflammatory and Immune Response After High Intensity Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marinova Pty Ltd (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network); University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: M01-21-01-T0011; NCT05181410 (obsolete NCT alias)
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Inflammatory Response
MeSH Terms: interventions — fucoidan

STUDY DESIGN:
Intervention Model Description: This is a prospective, double-blinded, placebo-controlled, cross-over design study. Participants will be randomized to one of the two SP sequences [either FMAS (2 weeks) → washout (1 week) → IPC (2 weeks): sequence A, or IPC (2 weeks) → washout (1 week) → FMAS (2 weeks): sequence B]. Each participant will act as their own control due to the cross-over design of the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both subjects and study research team will not be aware of their assigned conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fucoidan (Experimental): Fucoidan in Capsule
  Intervention: Dietary Supplement: Probiotic
  Interventions: Dietary Supplement: Fucoidan 500mg
- Placebo (Placebo Comparator): Non active ingredients in a capsule
  Intervention: Other: Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fucoidan 500mg — 1 capsule to be taken twice daily with food (morning and evening).
  Arms: Fucoidan
Dietary Supplement: Placebo — 1 capsule to be taken twice daily with food (morning and evening).
  Arms: Placebo

SUMMARY:
This double-blinded, randomized, placebo-controlled, cross-over study is designed to evaluate the potential effects of a fucoidan supplement on the inflammatory and immune responses following high intensity exercise.

DETAILED DESCRIPTION:
Inflammation is an innate immune response to tissue damage as a means of increasing blood flow to a specific area to facilitate repair, and is associated with the movement of fluid, plasma proteins, and immune cells from the circulation to the site of injury. The inflammatory process is initiated by cytokines which attract specific immune cells, such as monocytes, lymphocytes, neutrophils, and eosinophils, to the damaged tissue. Chronic exercise has been found to reduce inflammation and bolster immune system function; however, acute exercise has been shown to increase inflammatory response. Cytokine secretion and concentrations as well as leukocyte activation following exercise appear to increase in proportion to exercise intensity. Therefore, on an acute basis, high intensity exercise may cause immunosuppression and increased inflammation. High degrees of muscle damage and inflammation post-exercise result in decrements in muscle strength and range of motion, increased delayed onset muscle soreness (DOMS) and swelling, as well as the efflux of myocellular proteins and enzymes, including creatine kinase (CK). Therefore, post-exercise nutritional supplementation for individuals participating in high intensity exercise may be beneficial to modulate exercise-associated immune function and reduce inflammation.

Fucoidans are fucose-rich sulfated carbohydrates found in brown marine algae and have been shown to play a role in immune modulation as well as inflammation. In fact, fucoidans have been shown to inhibit neutrophil infiltration and attenuate levels of pro-inflammatory cytokines. More research is warranted to determine the effects of supplementation with fucoidans to reduce inflammation following high intensity exercise. Therefore, this double-blinded, randomized, placebo-controlled, cross-over design study will be conducted to further understand these effects.

ELIGIBILITY:
Inclusion Criteria:

1. Fully vaccinated against COVID-19 (participant has received their final dose at least one month prior to the screening visit).
2. Individuals who regularly exercise as per physical activity guidelines for Americans10 [structured exercise for a minimum of 150 cumulative minutes per week (low end) to 500 cumulative minutes of exercise per week (high-end)] and willing to maintain the same level of physical activity throughout the study period.
3. Healthy individuals between 18 to 40 years of age (inclusive).
4. Individuals with BMI in the range of 18.5-34.9 (inclusive).
5. Good health as determined by medical history and cleared for exercise as assessed by the PI.
6. Male and female participants of reproductive potential should be willing to use double-barrier to avoid pregnancy and sexually transmitted infection (STI) during the study period.
7. Provide signed and dated informed consent form.
8. Willing and able to comply with the protocol.

Exclusion Criteria:

1. Participants with existing musculoskeletal injuries that would prevent full participation.
2. History of clinically significant cardiovascular, respiratory, renal, cerebrovascular, metabolic, pulmonary, gastrointestinal, neurological, hematological, autoimmune, lymphatic, psychiatric, hepatobiliary, or endocrine disorders, including individuals with Type I or Type II diabetes, or other clinically significant medical condition that, in the opinion of the PI, may preclude safe study participation.
3. Females who are pregnant, lactating, or planning on becoming pregnant during the course of the study.
4. Participants using blood thinning medications or supplements.
5. Participants having a known sensitivity or allergy to any of the study products or their excipients.
6. Participating or has participated in another research study in which another study product has been consumed within 30 days prior to the study screening visit.
7. Participants with current or past medical history of long-term COVID-19 symptoms (remained symptomatic for at least 2 weeks or more).
8. Professional athletes, collegiate athletes, competitive body builders, or those who compete at the elite category within their sport.
9. Participant having any condition or abnormality that, in the opinion of the investigator, would compromise the safety of the participant or the quality of the study data.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in CBC panel | After 14 days of supplementation
  Changes in CBC panel (absolute counts of Neutrophils, Lymphocytes, Monocytes, Eosinophils, and Basophils) compared between two study arms to determine if the TP has an impact compared to placebo
Changes in interleukin-6 | After 14 days of supplementation
  To determine if the TP has an impact on interleukin-6 compared to placebo
Changes in interleukin-1B | After 14 days of supplementation
  To determine if the TP has an impact on interleukin-1B compared to placebo
Changes in interleukin-10 | After 14 days of supplementation
  To determine if the TP has an impact on interleukin-10 compared to placebo
Changes in T cell | After 14 days of supplementation
  Monitor changes in T cell subset CD4 and CD8 for TP compared to placebo
Changes in B cell | After 14 days of supplementation
  Monitor changes in B cell subset CD4 and CD8 for TP compared to placebo

SECONDARY OUTCOMES:
Safety Outcome Measures | After 14 days of supplementation
  Adverse events monitoring during the course of study to compare the safety of the TP compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Bridget McFadden, Principal Investigator — Principal Investigator
Locations (1):
- University of South Carolina Sport Science Lab, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No